CLINICAL TRIAL: NCT01555268
Title: A Phase lb Study of the Safety, Feasibility, and Pharmacokinetics of AMG 386 Alone and in Combination With Low Dose Cytarabine in Acute Myeloid Leukemia (AML) Patients
Brief Title: Trebananib With or Without Low-Dose Cytarabine in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 186010; NCI-2011-02979 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-16; First posted 2012-03-15 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — trebananib; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (trebananib) (Experimental): Patients receive trebananib IV over 30-60 minutes on days 1, 8, 15, and 22.
  Interventions: Biological: trebananib; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm B (trebananib, cytarabine) (Experimental): Patients receive trebananib as in Arm A. Patients also receive cytarabine SC BID on days 1-14 of course 1 and days 1-7 of subsequent courses.
  Interventions: Biological: trebananib; Drug: cytarabine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: trebananib — Given IV
  Other Names: AMG 386; AMG386
Drug: cytarabine — Given SC
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
  Arms: Arm B (trebananib, cytarabine)
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and the best dose of trebananib when given together with or without low-dose cytarabine in treating patients with acute myeloid leukemia (AML). Trebananib may stop the growth of AML by blocking blood flow to the cancer. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving trebananib together with cytarabine may be an effective treatment for patients with AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety, tolerability, and pharmacokinetic (PK) and pharmacodynamic (PD) profile of AMG 386 (trebananib) when administered alone and in combination with low-dose cytarabine in adult patients with: untreated AML considered ineligible for standard induction chemotherapy; refractory and/or relapsed AML following at least one cycle of prior therapy who are not currently eligible for stem cell transplantation.

SECONDARY OBJECTIVES:

I. To evaluate clinical responses in AML patients following AMG 386 therapy alone or in combination with low-dose cytarabine therapy.

II. To characterize the biological changes occurring in AML patients treated with AMG 386 alone or in combination with low-dose cytarabine, specifically: alteration in angiopoietin (Ang)1, Ang2, Tie2, vascular endothelial growth factor (VEGF), and VEGF receptor (VEGFR) expression; changes in bone marrow vascularization and hypoxia; changes in gene and/or micro ribonucleic acid (microRNA) expression; PK/PD modeling to characterize the time course of AMG 386 concentrations in relation to target inhibition and hematological response.

III. To determine whether the above biological changes correlate with and/or predict for clinical response in AML patients treated on this study.

OUTLINE: This is a dose-escalation study of trebananib. Patients are assigned to 1 of 2 treatment arms.

ARM A: Patients receive trebananib intravenously (IV) over 30-60 minutes on days 1, 8, 15, and 22.

ARM B: Patients receive trebananib as in Arm A. Patients also receive cytarabine subcutaneously (SC) twice daily (BID) on days 1-14 of course 1 and days 1-7 of each subsequent course.

In both arms, treatment repeats every 28 days* for up to 12 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Course 1 is 35 days.

After completion of study treatment, patients are followed up for 30 days, every month for 1 year, every 3 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML as defined by the World Health Organization (excluding acute promyelocytic leukemia and chronic myeloid leukemia- blast/accelerated phase) in an adult patient

  * Patients with newly diagnosed untreated AML for whom the treatment of choice is low-intensity therapy by investigator assessment or who has declined intensive induction therapy recommended by the investigator OR
  * Patients with refractory or relapsed AML following at least one prior treatment course who are not currently considered eligible for stem cell transplantation at the time of screening due to non-optimal AML disease control, lack of suitable transplantation donor, failure to meet other transplantation criteria, or refusal to undergo transplantation
* Eastern Cooperative Oncology Group (ECOG) status 0-2 (ECOG 3 is excluded)
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN)
* Creatinine clearance > 40ml/min per 24 hour urine collection or calculated according to the Cockcroft-Gault formula
* Urinary protein quantitative value of less than 30mg/dL in urine analysis or less than 1+ on dipstick, unless quantitative protein is < 1000mg in a 24 hour urine sample
* Partial thromboplastin time (PTT) or activated (aPTT) =< 1.5 x ULN per institution laboratory range and international normalized ratio (INR) =< 1.5
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Individuals of childbearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment

Exclusion Criteria:

* History of central nervous system involvement with leukemia
* History of venous or arterial thromboembolism within 12 months prior to enrollment
* History of clinically significant bleeding within 6 months of enrollment
* Unresolved toxicities from prior systemic therapies that are Common Terminology Criteria for Adverse Events (CTCAE) version 4 >= Grade 2 in severity except alopecia excluding hematological toxicities attributable to underlying disease
* Currently or previously treated with AMG 386, or other molecules that inhibit the angiopoietins or Tie2 receptor
* Current or within 30 days prior to enrollment treatment with immune modulators such as systemic cyclosporine or tacrolimus
* Has not yet completed a 14 day washout period for any previous anti-cancer systemic therapies (30 days for prior bevacizumab) with the exception of hydroxyurea or leukapheresis for uncontrolled leukocytosis
* Enrolled in or has not yet completed at least 14 days since ending other investigational device or drug trials, or currently receiving other investigational treatments
* Clinically significant cardiovascular disease within 12 months prior to enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication or placement of percutaneous transluminal coronary angioplasty/stent
* Major surgery within 28 days prior to enrollment or still recovering from prior surgery
* Minor surgical procedures, placement of tunneled central venous access device within 3 days prior to enrollment
* Uncontrolled hypertension as defined as diastolic > 90mmHg OR systolic > 140mmHg; the use of anti-hypertensive medication to control hypertension is permitted
* Non-healing wound, ulcer (including gastrointestinal) or fracture
* Active uncontrolled infection, including human immunodeficiency virus (HIV) and active hepatitis infection
* Subject not consenting to the use of highly effective contraceptive, e.g., double barrier method (i.e., condom plus diaphragm) precautions during the course of the study and for 6 months after administration of the last study medication
* Subject has known sensitivity to any of the products to be administered during dosing
* History of allergic reactions to bacterially produced proteins
* Subject has previously been enrolled onto this study
* Subject will not be available for follow-up assessment
* Pregnant or nursing female patients
* Active second malignancy other than AML which is not in remission and/or for which the patient is currently receiving treatment
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Any condition which in the investigator's opinion makes the patient an unsuitable candidate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2013-09-24 (Actual); Study Completion 2016-08-03 (Actual)

PRIMARY OUTCOMES:
Safety of trebananib when administered alone and in combination with low-dose cytarabine measured by number of participants with toxicities according to CTCAE | Up to 30 days after the last dose of study drug
  Adverse events will be tabulated overall and by arm.
PK/PD profile of trebananib when administered alone | Days 1, 3-5, 7, 8, 22, 24-26, and 29 of course 1
  A population PK/PD model will be developed to characterize the time course of AMG 386 concentrations in relation to target inhibition and hematological response. Model-predicted PK parameters will be generated, such as individual areas-under-the-curve (AUCs) and Cmax for AMG 386, to correlate with targeted biomarkers, such as Ang1, and Ang2, and VEGF as well as leukocyte count.
PK/PD profile of trebananib when administered in combination with low-dose cytarabine | Days 1 and 7 of course 1
  A population PK/PD model will be developed to characterize the time course of AMG 386 concentrations in relation to target inhibition and hematological response. Model-predicted PK parameters will be generated, such as individual AUCs and Cmax for AMG 386, to correlate with targeted biomarkers, such as Ang1, and Ang2, and VEGF as well as leukocyte count.

SECONDARY OUTCOMES:
Clinical response in AML patients following trebananib therapy alone or given in combination with low-dose cytarabine therapy | Up to 5 years
Alterations in Ang1, Ang2, Tie2, VEGF, and VEGFR expression | Up to 30 days post-treatment
  Identified by flow cytometric analysis of peripheral blood and marrow aspirate cells.
Changes in bone marrow vascularization and hypoxia | Baseline up to 30 days post-treatment
  Bone marrow vascularization will be assessed by cluster of differentiation (CD)31+ and/or CD34 microvessel staining as well as VEGF-A expression and hypoxia using hypoxia-inducible factor (HIF)-1alpha and/or CAIX immunohistochemistry.
Changes in gene and/or microRNA expression | Baseline up to 30 days post-treatment
  Microarray profiling for all human microRNAs will be performed on stored leukemia marrow cells and confirmed by real time-polymerase chain reaction (Q-PCR) analysis for specific microRNAs of interest.
Characterization of time course of trebananib concentrations in relation to target inhibition and clinical response using PK/PD modeling | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Wang, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York